CLINICAL TRIAL: NCT05900362
Title: Feasibility and Success Trial of Remote Patient Monitoring in Heart Failure
Acronym: FAST-RPM-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Luke's Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2021-03-28; First posted 2023-06-12 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Interventional (Experimental): All patients receive the VitalCare platform with a tablet computer, an Eko Duo device, a weight scale, a blood pressure cuff, a pulse oximeter
  Interventions: Device: VitalCare Platform

INTERVENTIONS:
Device: VitalCare Platform — All participants will receive an VitalCare platform with tablet, Eko Duo with capability to record heart/lung sounds, blood pressure cuff, pulse oximetry and digital scale

SUMMARY:
Previous research has investigated the use of remote patient monitoring in various clinical contexts, however there has not been a clinical trial examining use of the VitalCare platform for ambulatory management of heart failure. This trial will serve as a pilot study examining the feasibility of use of the VitalCare platform for ambulatory heart failure management and examine the effect of remote patient monitoring on patient engagement. To the investigators' knowledge, this will be the first study examining the effect of remote patient monitoring with the VitalCare platform on heart failure clinical outcomes, such as hospitalization for heart failure exacerbations and emergency room visits for heart failure.

DETAILED DESCRIPTION:
The next step in determining the role of remote patient monitoring in the management of patients with heart failure is to better understand which patients are most likely to benefit from a more intensive outpatient management or simply conservative management. The subject population is patients with mild HFrEF or HFpEF who are prone to readmission. This patient population does not have implanted devices to supply objective data to evaluate patient's volume status and therefore can be challenging to manage on an outpatient basis. By providing regular data on weight, blood pressure, pulse oximetry, electrocardiogram and heart/lung sounds that is reviewed on a monthly basis, this may allow a clinician greater insight into their patient's clinical status and allow for a more accurate and timely intervention to prevent clinical deterioration. Furthermore, this should enhance patient engagement with their own health as well as with their healthcare provider. This study would significantly add to the current knowledge of management of heart failure in an ambulatory patient population without implanted devices.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of heart failure
* New York Heart Association Class II or III congestive HF symptoms
* Admission to hospital within 12 months for symptomatic heart failure.
* Own a smartphone or tablet or comfortable with using one
* English as primary language
* Able to provide informed consent

Exclusion Criteria:

* Left Ventricular Ejection Fraction < 35%
* Implanted cardiac device (permanent pacemaker (PPM), implantable cardioverter defibrillator (ICD), chronic resynchronization therapy (CRT), implantable loop recorder (ILR))
* CardioMEMS
* Left ventricular assist device (LVAD)
* NYHA Class I or IV congestive HF symptoms
* Listed for cardiac transplant
* Pregnant at time enrollment
* End-stage renal disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Compliance with monitoring protocol | 6 month
  Actual rate of completed patient data transmissions is greater than or equal to 60% of the expected rate of patient data transmissions (BP, HR, Weight, EKG)

SECONDARY OUTCOMES:
Patient engagement as measured by Patient Activation Measure | 6 months
  Patient engagement as measured by the Patient Activation Measure will increase by 1 or more points from baseline to 6 months. The PAM score ranges from 1 to 100 corresponding to 1 of 4 levels of patient engagement. Higher numbers correlate with greater patient engagement.
Heart failure hospitalizations, emergency room visits for Heart Failure as compared to prior to trial enrollment | 6 month
  Patients who undergo remote patient monitoring via the VitalCare platform will have a lower rate of hospitalization for heart failure and lower rate of emergency room presentation for heart failure symptoms as compared to previous rate of heart failure hospitalization and emergency room presentations for heart failure symptoms for the 6 months prior to trial enrollment

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Saint Luke's Hospital of Kansas City, Kansas City, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Saint Luke's North Hospital, Kansas City, Missouri
  - Saint Luke's East Hospital, Lee's Summit, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Mid 2021
Access Criteria: Contact PI